CLINICAL TRIAL: NCT01834664
Title: Safety and Efficacy of Bone Marrow Derived Autologous Cells for the Treatment of Cerebral Palsy in Subjects Above Years (BMACCP) .It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Safety and Efficacy of Bone Marrow Derived Autologous Cells Treatment of Cerebral Palsy in Subjects Above 15 Years
Acronym: BMACCP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, CO-Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00109
Record Dates: First submitted 2013-04-08; First posted 2013-04-18 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Ataxic Infantile Cerebral Palsy
Keywords: Ataxic Infantile Cerebral Palsy stem cell therapy
MeSH Terms: conditions — Cerebral Palsy, Ataxic, Autosomal Recessive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STEM CELL (Other): Transfer of autologous stem cell [MNCs ]intrathecally
  Interventions: Biological: stem cell (MNCs )

INTERVENTIONS:
Biological: stem cell (MNCs ) — Intra thecal transplantation of autologous stem cell [MNCs ]Per dose at the interval
  Other Names: Intra thecal autologous stem cell MNCs

SUMMARY:
This Study is Single arm, Single Centre trial to study the safety and efficacy of bone marrow derived autologous mononuclear cells (100 millions per dose)study enrollment duration 36 months sample size 100 patients should be treated (above 15 years of age) with cerebral palsy in India. Primary outcome measures are improvement in walking ability and kinetic gait pattern.

DETAILED DESCRIPTION:
Cerebral Palsy is commonest cause of Disability in India and south East Asia. This Study is devised to quantify the safety and efficacy of bone marrow derived autologous mononuclear cells(100 millions per dose)study enrolment duration 36 months sample size 100 patients should be treated (above 15 years of age) with cerebral palsy, in India. Primary outcome measures are improvement in walking ability and kinetic gait pattern as per as various clinical scales and also changes in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged above 15 years with a diagnosis of Cerebral Palsy. Regional Nerve damage as shown by Magnetic Resonance Imaging(MRI)
* Patient suffer from cerebral palsy due to prenatal and postnatal cause,
* Willing to undergoing Bone Marrow derived autologous stem cell therapy.
* Able to Comprehend and give written informed consent form for the study
* willing to come to the hospital for follow up visits as per the protocol requirements

Exclusion Criteria:

* History of meningitis,meningoencephalitis , epilepsy or life threatening allergic or immune -mediated reaction
* Hemodynamically unstable patients
* history of or concurrent autoimmune disease or acute episode if Guillain- barre syndrome
* peripheral Muscular dystrophy

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in muscle rigidity using Ash worth scale | 6 Months

SECONDARY OUTCOMES:
Improvement in dysregulated phospholipid Metabolism | 6 months
Improvement in walking ability and kinetic gait Pattern | 6 Months
Improvement in overall motor control using oxford scale | 6 Months
Improvement in orbitoFrontal-amygdala circuit and self-regulation of social -emotional behaviour | 6 month
Improvement in motor-linked implicit learning | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, M.S, Principal Investigator — CHAITANYA HOSPITAL
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India